CLINICAL TRIAL: NCT02465359
Title: A Study of Subcutaneous Immunoglobulin as Chronic Treatment for Patients With Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: Subcutaneous Immunoglobulin for Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Acronym: SCIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00016957
Record Dates: First submitted 2014-12-12; First posted 2015-06-08 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — gamma-Globulins; Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immune globulin subcutaneous (Human) (Experimental): lmmune Globulin Subcutaneous(Human) 20% Liquid (Hizentra) will be given weekly
  Interventions: Drug: Immune Globulin Subcutaneous (Human)

INTERVENTIONS:
Drug: Immune Globulin Subcutaneous (Human) — Patients who have CIDP and are on IVIG will be allowed in the study to try subcutaneous immune Globulin (SCIG) as part of an open label study.
  Other Names: Hizentra

SUMMARY:
The investigators are using self administered subcutaneous immunoglobulin (SCIG) in patients with CIDP who require Intravenous immunoglobulin (IVIG). Safety, efficacy, and patient satisfaction will be examined.

DETAILED DESCRIPTION:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is an autoimmune neurological disorder that causes limb weakness and numbness. Many patients require immunosuppressants and plasma exchange (PLEX) to control their symptoms. Intravenous immunoglobulin (IVIG) is also an effective treatment (Hughes et al, 2006 & 2008; Hughes, 2009; Cocito et al, 2010), and the American Academy of Neurology (AAN) guideline recommended that it should be offered in the long-term treatment of CIDP (Patwa et al, 2012). While effective, IVIG causes systemic side effects in about 5% of patients. These side effects include rash, pruritus, myalgia, fever, chills, headache, low back pain, nausea, vomiting, changes in blood pressure or heart rate, renal failure, and aseptic meningitis (Berger, 2008). For many patients who are chronically treated with IVIG, venous access may be a problem over time. An alternative is the subcutaneous (SC) route, which has been in use since 1980 for primary immune deficiency disorders and is the treatment of choice for this condition in Scandinavia and England (Radinsky et al, 2003). As compared to intravenous (IV) route, SC route maintains higher trough levels of immunoglobulins, increases patient independence, reduces systemic side-effects, and is better tolerated in those who are pregnant or sensitized to Immunoglobulin A (IgA) (Radinsky et al, 2003). In a review of side effects associated with 33,168 SCIG infusions, no severe or anaphylactoid reactions occurred (Gardulf et al, 1995). Patients can self-administer medication, and hence, overall cost may be reduced. A retrospective study of 28 children with primary immunodeficiency in Canada showed that the mean difference in costs between IVIG and SCIG during the study period (1 year on IVIG and 1 year on SCIG) was $4,346 in favor of SCIG (Ducruet et al, 2011). A US$10,100 reduction in cost per year per patient associated with SCIG use was also reported by Gardulf et al (1995) in Sweden. Disadvantages of SCIG include more frequent infusions and local reactions at sites of infusion (transient swelling, soreness, redness, induration, local heat, and itching) in about 1% of patients.

ELIGIBILITY:
Inclusion Criteria:

To qualify, a patient must have CIDP and persistence of significant symptoms (having 2 or more of the following):

* Weakness in any limb,
* Motor fatigue significant to interfere with activities of daily living (ADL) or work,
* Paresthesia of sufficient severity to require a medication,
* Sensory impairment,
* Walking impairment,

AND requires IVIG to control symptoms.

Exclusion Criteria:

1. Thrombocytopenia or other bleeding disorders,
2. Anticoagulation therapy,
3. Severe or anaphylactoid reactions to IVIG,
4. Cancer,
5. Pregnancy,
6. Breast-feeding,
7. Renal insufficiency or failure,
8. Congestive heart failure,
9. Psychiatric illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuan Vu, MD, Principal Investigator — University of South Florida
Locations (1):
- USF Dept of Neurology, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Immune Globulin Subcutaneous (Human): lmmune Globulin Subcutaneous(Human) 20% Liquid (Hizentra) will be given weekly
  Immune Globulin Subcutaneous (Human): Patients who have CIDP and are on intravenous immunoglobulin (IVIG) will be allowed in the study to try subcutaneous immune Globulin (SCIG) as part of an open label study.
Period: Overall Study
Arm/Group | Immune Globulin Subcutaneous (Human)
Started | 15
Completed | 12
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15
Duration of IVIg use before SCIg (months) [Mean (Standard Deviation); unit: Months] | 25.8 (24.01)

OUTCOME MEASURES:

1. Primary Outcome: Relapse of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Symptoms
Description: This outcome measure, referred to as the relapse of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) symptoms, is a measure of how many participants experiences CIDP symptoms causing them to withdraw prematurely from the study. This is a count of participant withdrawals compared to the number of participants who completed the study.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
Participants
  withdrew prematurely | 3
  completed study | 12

2. Secondary Outcome: Mean Change in Short Form 36 (SF-36) Domain: Physical Functioning Between Week 24 and Screening
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to physical functioning is shown, listed as the mean change from screening to 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0 [-0.12 to 0.12]

3. Secondary Outcome: Mean Change in Inflammatory Rasch-built Overall Disability Scale (I-RODS) From Screening to Week 24
Description: The Inflammatory Rasch-built Overall Disability Scale (I-RODS) is an instrument answered by the patient to assess overall disability through assessing activity and social participation limitations in patients with inflammatory neuropathies. It is a 24-item scale, with each item representing a common, daily activity. The patient assigns a score between 0 and 2 to each item as follows:
  0 = impossible to perform
  1. = performed with difficulty
  2. = easily performed
  The total raw score on the I-RODS (0-48 max) is transformed to a final score (0-100), with a lower score indicating worse outcomes. Here the outcome measure is the mean change between screening and week 24, as calculated from transformed total I-RODS score. A negative change between week 24 and screening, or a reduction in I-RODS score, indicates a worsening of the patient's perceived daily functioning, as measured by the I-RODS.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 14
units on a scale | -1.5 [-4.6 to 1.6]

4. Secondary Outcome: Mean Change in Chronic Acquired Polyneuropathy Patient-Reported Index (CAP-PRI) Between Week 24 and Screening
Description: The Chronic Acquired Polyneuropathy Patient-Reported Index (CAP-PRI) is used to evaluate quality of life in patients with polyneuropathy. The scale consists of 15 items, resulting in a single-score with 4 life domains (physical, social, pain and emotional well-being). Each item assessed is scored 0-2 (0= not at all, 1 = a little bit, 2 = a lot). Max score possible is 30 with a higher score indicating worse outcomes.
  This outcome measure was evaluated at screening and week 24 by determining the mean change between these two time points. A negative score would indicate an improvement as perceived by the participant.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
units on a scale | -4.3 [-7.7 to -0.9]

5. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) is used to assess the patient's treatment satisfaction with intravenous immune globulin (IVIg) compared to the use of subcutaneous immune globulin (SCIg). There are 14 items and the TSQM addresses four domains: effectiveness, side effects, convenience, and global satisfaction. Questions are scored from one (least satisfied) to five or seven (most satisfied), with the exception of item 4 relating to side effects (scored yes/no, 1 or 0, respectively). Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100. Higher scores indicate higher treatment satisfaction.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 11
units on a scale | 10.3 [4.3 to 16.2]

6. Secondary Outcome: Mean Change in Short Form 36 Domain: Role Limitations-physical Between Screening and Week 24
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "role limitations-physical" is shown, listed as the mean change between screening to 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0.24 [0.03 to 0.46]

7. Secondary Outcome: Mean Change in Short Form 36 Domain: Role Limitations - Emotional (Between Week 24 and Screening)
Description: The short form 36 (SF-36) measure health status of patients. Per Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "role limitations-emotional" is shown, listed as the mean change from screening to 24 weeks.
  A negative value for this measure indicates a worsening of role limitations related to emotional health.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | -0.01 [-0.27 to 0.24]

8. Secondary Outcome: Mean Change in Short Form 36 Domain: Energy/Fatigue Between Screening and Week 24
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "energy/fatigue" is shown, listed as the mean change between screening and 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0.09 [0.00 to 0.18]

9. Secondary Outcome: Mean Change in Short Form 36 Domain: Emotional Well-being Between Screening and 24 Weeks
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "emotional well-being" is shown, listed as the mean change between screening and 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0.03 [-0.04 to 0.09]

10. Secondary Outcome: Mean Change in Short Form 36 Domain: Social Functioning Between Screening and Week 24
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "social functioning" is shown, listed as the mean change between screening and 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0.06 [-0.07 to 0.19]

11. Secondary Outcome: Mean Change in Short Form 36 Domain: Pain Between Screening and 24 Weeks
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "pain" is shown, listed as the mean change between screening and 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0.08 [0.00 to 0.16]

12. Secondary Outcome: Mean Change in Short Form 36 Domain "General Health" Between Screening and Week 24
Description: The short form 36 (SF-36) is a health status profile designed to measure health status and outcomes of patients. Per the paper from Burholt and Nash (2011) scoring and domains are as follows:" The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health." For this particular outcome measure, only the domain pertaining to "general health" is shown, listed as the mean change between screening and 24 weeks.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
score on a scale | 0.01 [-0.07 to 0.10]

13. Secondary Outcome: Mean Change in Limb Motor Strength Testing (LMST) Over 24 Weeks
Description: LMST is a discrete variable that tests muscle strength in upper and lower limbs. It is a sum of the strength of 16 muscle groups tested at a given time point. LMST is measured and reported in pounds (lbs). For this outcome measure, the mean change, in pounds, between screening and week 24 LMST is reported.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
pounds | 5.6 [2.3 to 8.9]

14. Secondary Outcome: Mean Change in Timed 25-foot Walk (T25-FW) Between Screening and Week 24
Description: The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk. A lower time indicates greater mobility and leg performance, thus suggesting better outcomes. Time is measured in seconds. This outcome is the mean change between timed 25 foot walk times between screening and week 24.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Immune Globulin Subcutaneous (Human)
Number analyzed (Participants) | 15
seconds | -1.0 [-2.9 to 0.8]

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Definitions do not differ to ClinicalTrials.gov adverse event definitions.
Arm/Group | Immune Globulin Subcutaneous (Human)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 13/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immune Globulin Subcutaneous (Human) (N=15)
Pain at infusion site (General disorders) | 13
Transient swelling at site of infusion (General disorders) | 12
Redness at site of infusion (General disorders) | 11
Induration at site of infusion (General disorders) | 7
Itching at site of infusion (General disorders) | 7
Numbness (General disorders) | 5
Bruising at site of infusion (General disorders) | 5
Increased Exhaustion (General disorders) | 4
Hedache/Migrane (Nervous system disorders) | 4
Local heat at site of infusion (Skin and subcutaneous tissue disorders) | 3
Increased weakness (Musculoskeletal and connective tissue disorders) | 3
Tingling sensation (Skin and subcutaneous tissue disorders) | 3
Burning sensation at site of infusion (Skin and subcutaneous tissue disorders) | 3
Fever (General disorders) | 2
Pain in the extremities (Musculoskeletal and connective tissue disorders) | 2
Fell/fainted (General disorders) | 2
Generalized itching (Skin and subcutaneous tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Stabbing Pain (General disorders) | 1
Backache (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Twitching (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
CIDP exacerbation (Nervous system disorders) | 1
Heavy legs (General disorders) | 1
Bleeding at site of infusion (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Stiffness (Musculoskeletal and connective tissue disorders) | 1
Eyes burning (Eye disorders) | 1
Shingles (General disorders) | 1
Severe hip osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
Small, open-label trial; lacks immunoglobulin G (IgG)-dependency test; predictors of poor QOL were not substratified during analysis of the primary and secondary endpoints; lack of baseline IVIg observation period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT02465359/Prot_SAP_000.pdf